CLINICAL TRIAL: NCT05451303
Title: Detection of Oral and Throat Cancers Using Saliva Metatranscriptomic Analysis
Brief Title: Detection of Oral and Throat Cancers Using OralViome Cancer Testing System
Status: Recruiting | Type: Observational
Sponsor: Viome (Industry)
Collaborators: New York Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: V300
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Oral Squamous Cell Carcinoma; Oropharynx Squamous Cell Carcinoma; Premalignant Lesion
Keywords: Viome; oral cancer; detection; OSCC; OPMD-B; OPMD-PM; OPMD; OPV; Tobacco; HPV
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Oral Squamous Cell Carcinoma (OSCC): OSCC case cohort will consist of patients with Oral Squamous Cell Carcinoma (all stages, locations), recruited from secondary care.
  Interventions: Device: OralViome Cancer Testing System
- OroPharyngeal Cancer (OPC): OPC case cohort will consist of patients with OroPharyngeal cancer (all stages, locations), recruited from secondary care.
  Interventions: Device: OralViome Cancer Testing System
- Oral Potentially Malignant Disease (OPMD): OPMD cohort will consist of patients with both potential malignancies or benign conditions including, but not limited to:
  * Dysplasia
  * Hyperplasia
  * Leukoplakia
  * Erythroplasia
  * Lichenoid lesions
  * Actinic Keratosis
  * Lichenoid reaction
  * Aphthous ulcer/ Canker Sores
  * Gingival enlargement (side effect)
  * Lichen planus
  * Keratosis
  * Inflammatory reaction
  * Cheek bites
  Interventions: Device: OralViome Cancer Testing System
- Cancer-free: Cancer free control cohort will be matched with cases. Participants will be recruited following clinical adjudication with self-reported confirmation of no cancer and from primary care facilities.
  Interventions: Device: OralViome Cancer Testing System

INTERVENTIONS:
Device: OralViome Cancer Testing System — The OralViome Cancer Testing System is intended for the screening of Oral Squamous Cell Carcinoma (OSCC) and Oropharyngeal cancer (OPC). The system consists of the OralViome Saliva Collection and Transport Kit, the Viome laboratory process for metatranscriptomics, and the Viome analytical software that detects an RNA expression signature within a saliva sample.

SUMMARY:
To evaluate the design, safety and efficacy of OralViome Cancer Testing system in the early detection of Oral and Throat Cancers using saliva metatranscriptomic analysis. This study will recruit only at existing clinical sites and will NOT use any additional clinical sites.

DETAILED DESCRIPTION:
This is an observational study evaluating the design, safety and efficacy of OralViome Cancer Testing system in the early detection of Oral and Throat Cancers using saliva metatranscriptomic.

A total of 475 participants will be recruited, including 4 different cohorts: 1) cancer free patients, 2) patients with Oral Potentially Malignant Disease (OPMD), 3) patients with Oral Squamous Cell Carcinoma (OSCC), and 4) patients with OroPharyngeal Cancer (OPC). OSCC and OPC participants will be recruited from secondary care facilities, OPMD and cancer free participants will be recruited from primary care facilities.

Participants will complete health questionnaires and collect saliva samples using at home/ in clinic kits provided by Viome. The duration of study participation will be 1 clinic visit for cancer free participants, and up to 1 year for those with OSCC/OPC/OPMD.

ELIGIBILITY:
Inclusion Criteria

* Signed Informed Consent obtained
* 18 years and older
* At a high risk of developing oral or throat cancer based on clinician's discretion

Exclusion Criteria

* Pregnancy
* Use of fertility enhancing medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited into one of four cohorts, OSCC, OPC, OPMD, or cancer free cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 475 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the detection or not of OSCC or OPC | 1 year
  The test results will be compared against the definitive diagnosis by the physician.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Julian, PhD, Principal Investigator — Viome
Locations (1):
- NYMC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No